CLINICAL TRIAL: NCT01670617
Title: A Stratified, Post-Market Study of DeNovo NT for the Treatment of Femoral and Patellar Articular Cartilage Lesions of the Knee
Brief Title: DeNovo NT Natural Tissue Graft Stratified Knee Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zimmer Orthobiologics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSU2011-03B
Record Dates: First submitted 2012-08-08; First posted 2012-08-22 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2016-12

CONDITIONS: Defect of Articular Cartilage; Knee Injuries
MeSH Terms: conditions — Knee Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DeNovo NT Graft (Other): DeNovo NT Graft stratified by lesion location - femur or patella
  Interventions: Other: Particulated Juvenile Articular Cartilage

INTERVENTIONS:
Other: Particulated Juvenile Articular Cartilage — Treatment of articular cartilage defects up to 7.5 cm2
  Other Names: DeNovo NT Natural Tissue Graft

SUMMARY:
The purpose of this study is to evaluate the long-term relief of pain and return to function for patients receiving DeNovo NT for cartilage lesions in the knee. DeNovo NT is a marketed product and has been used in more than 7,500 patients over the last 7 years.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Voluntary signature of the IRB approved Informed Consent,
2. Male or female subjects between the ages of 18 to 55 years,
3. If female: Actively practicing a contraception method and willing to continue for a minimum of 1 year postoperatively, practicing abstinence and willing to continue for a minimum of 1 year postoperatively, or sterile
4. One or two contained lesion(s) of the femur or patella ≥ ICRS Grade 3 or OCD lesions with healed bone base with no loss of bone greater than 6mm
5. Has peripheral cartilage debridement to healthy cartilage that results in at least one lesion with an area of ≥ 2 cm2 and ≤ 7.5 cm2,
6. Lesion(s) to be treated must be contained/shouldered > 70% of the periphery,
7. Ligaments in the affected knee are stable,
8. Ipsilateral knee compartment has intact menisci
9. The contralateral knee is asymptomatic, stable, and fully functional,
10. Is refractory to conservative non-surgical management or minimal surgical intervention and ≥ 3 months from the start of either treatment,
11. Must record a response, at the preoperative study visit, of moderate to extreme pain for any one of the KOOS Pain Scale questions, P2 through P9.
12. Must be physically and mentally willing and able, in the Investigator's opinion at the time of enrollment, to be compliant with the protocol

EXCLUSION CRITERIA:

1. Clinical disease diagnosis of the indexed affected joint that includes

   * Osteoarthritis or avascular necrosis,
   * Rheumatoid arthritis, or history of septic or reactive arthritis,
   * Gout or a history of gout or pseudogout in the affected knee,
   * Bipolar articular cartilage involvement (or kissing lesions)
   * Has more than two clinically relevant chondral lesion(s) on the index knee,
   * Osteochondritis dissecans of the knee with significant bone loss
   * Associated damage to the underlying subchondral bone requiring bone graft,
   * Has well-defined subchondral cyst(s),
   * Has current or impending subchondral avascular necrosis,
2. History of secondary arthropathies (i.e., sickle cell disease, hemochromatosis, or autoimmune disease),
3. Uncontrolled diabetes,
4. Displays a high surgical risk due to unstable cardiac and/or pulmonary disease,
5. Has HIV or other immunodeficient state
6. Is at substantial risk for the need of organ transplantation
7. Is pregnant or breast-feeding,
8. Body Mass Index >35 (BMI=kg/m2),
9. Is participating concurrently in another clinical trial
10. Is receiving prescription pain medication other than NSAIDs or acetaminophen for conditions unrelated to the index knee condition, chronic use of anticoagulants, or taking corticosteroids,
11. Has a neuromuscular, neurosensory, or musculoskeletal deficiency that limits the ability to perform objective functional assessment of either knee,
12. Active joint infection or history of chronic joint infection at the surgical site,
13. Prior total meniscectomy of either knee,
14. Has severe patellofemoral malalignment/maltracking or patellar instability
15. Radiographically has >5 degrees of malalignment
16. Has received, within the past 3 months HA or cortisone injections in knee,
17. Has undergone prior tendon repair, meniscus repair, ligament repair or distal realignment/osteotomy surgery in the index knee, < 6 months prior to surgery,
18. Failed marrow stimulation or ACI treatment performed < 12-mo before baseline,
19. Index knee has been surgically treated for cartilage repair with OATs, mosaicplasty or osteochondral allograft,
20. Involves concomitant procedures in the affected knee with the exception of incidental loose body removal, debridement, synovectomy, retinacular release, and/or partial meniscectomy
21. Has contraindications for Magnetic Resonance Imaging (MRI),
22. Has an allergy to Polymyxin B sulfate or Bacitracin antibiotics,
23. Is receiving workman's compensation or currently involved in litigation relating to the index knee

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2012-03; Primary Completion 2018-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Improvement in KOOS scores | Between baseline and 24 months post surgery
  Improvement in Knee Injury and Osteoarthritis Outcomes Survey (KOOS) scores

SECONDARY OUTCOMES:
X-ray Evaluation | Preop, 12 months and 24 months post surgery
  X-ray evaluation of joint narrowing, and osteophyte and cyst formation
Incidence and time to reoperation/revision | 5 years
Mean IKDC Knee Examination grades | Annually to 5 years post surgery
MRI Evaluation | Preop, 12 Months and 24 Months post surgery
  Magnetic Resonance Observation of Cartilage Repair Tissue (MOCART) score
Incidence of adverse events | Annually to 5 years post surgery

CONTACTS AND LOCATIONS:
Locations (18):
- United States (16):
  - Kerlan Jobe Orthopaedics, Los Angeles, California
  - Naval Medical Center San Deigo, San Deigo, California
  - Colorado Orthopedic Consultants, Aurora, Colorado
  - Andrews Institute for Orthopaedics & Sports Medicine, Gulf Breeze, Florida
  - Emory Spine & Sports Medicine Center, Atlanta, Georgia
  - Tulane University Medical Center, New Orleans, Louisiana
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - TRIA Orthopaedic Center, Bloomington, Minnesota
  - Minnesota Orthopedic Sports Medicine Institute at Twin Cities Orthopedics, Edina, Minnesota
  - A.T. Still University of Health Sciences, Kirksville, Missouri
  - University Orthopaedic Associates, Somerset, New Jersey
  - New Mexico Orthopaedic Consultants, Albuquerque, New Mexico
  - Oregon Health & Science University, Portland, Oregon
  - San Antonio Military Medical Center, San Antonio, Texas
  - University of Virginia, Charlottesville, Virginia
  - Madigan Army Medical Center, Tacoma, Washington
- Canada (2):
  - Ottawa Hospital, Ottawa, Ontario
  - Women's College Hospital, Toronoto

REFERENCES:
- [Background] Farr J, Cole BJ, Sherman S, Karas V. Particulated articular cartilage: CAIS and DeNovo NT. J Knee Surg. 2012 Mar;25(1):23-9. doi: 10.1055/s-0031-1299652. PMID 22624244